CLINICAL TRIAL: NCT00004288
Title: Phase II Pilot Study of Olsalazine for Ankylosing Spondylitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: University of Rochester (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Treatment
Other Study IDs: 199/11716; URMC-44
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-01

CONDITIONS: Ankylosing Spondylitis
Keywords: ankylosing spondylitis; genetic diseases and dysmorphic syndromes; rare disease
MeSH Terms: conditions — Spondylitis, Ankylosing; Genetic Diseases, Inborn; Rare Diseases | interventions — olsalazine

INTERVENTIONS:
Drug: olsalazine

SUMMARY:
OBJECTIVES:

I. Assess the safety and efficacy of olsalazine, a dimer of 5-aminosalicylic acid, in men with ankylosing spondylitis unresponsive to nonsteroidal anti-inflammatory drugs and physiotherapy.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Patients are treated with daily olsalazine. The dose is increased each week until the protocol dose is reached.

Supplemental acetaminophen is allowed; nonsteroidal anti-inflammatory drugs continue unchanged. Concurrent sulfasalazine is prohibited.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Meets modified New York diagnostic criteria
* Active disease, i.e., morning stiffness for more than 30 minutes
* Failed or experienced nonlife-threatening reaction to prior sulfasalazine
* No significant hematologic, hepatic, or renal disease

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4
Dates: Start 1996-05; Study Completion 1999-12

CONTACTS AND LOCATIONS:
Overall Officials: Samuel H. Zwillich, Study Chair — University of Rochester